CLINICAL TRIAL: NCT02233244
Title: A Phase 1, Open-Label, Two-Period, Fixed-Sequence, Drug-Drug Interaction Study to Evaluate the Pharmacokinetics and Safety of CTX 4430 and Midazolam in Healthy Adult Subjects
Brief Title: Drug-Drug Interaction Study to Evaluate the Pharmacokinetics and Safety of CTX 4430 and Midazolam
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celtaxsys, Inc. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CTX-4430-DI-001
Record Dates: First submitted 2014-07-22; First posted 2014-09-08 (Estimated); Last update posted 2014-10-10 (Estimated); Status verified 2014-10

CONDITIONS: Healthy
Keywords: Drug Interaction
MeSH Terms: interventions — acebilustat; Midazolam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CTX-4430 and midazolam (Other): Midazolam 2 mg solution once, CTX-4430 100 mg tablet once per day for 7 days, Midazolam 2 mg solution once
  Interventions: Drug: CTX-4430; Drug: Midazolam

INTERVENTIONS:
Drug: CTX-4430
Drug: Midazolam

SUMMARY:
This drug-drug interaction study will assess the potential of CTX-4430 to induce CYP3A activity in healthy subjects.

The study hypothesis is that midazolam (a sensitive, widely used CYP3A4 substrate) blood levels will not change after treatment with CTX-4430.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult male or female, 18-55 years of age, inclusive at screening
* Continuous non-smoker who has not used nicotine-containing products for at least 3 months prior to the first dose
* Body Mass Index (BMI) ≥ 18.5 and ≤ 32.0 kg/m2 at screening
* Medically healthy with no clinically significant medical history, physical examination, laboratory profiles, vital signs or ECGs, as deemed by the PI
* For a female of childbearing potential: either be sexually inactive (true abstinence in line with the preferred and usual lifestyle of the subject) for 14 days prior to the first dose and throughout the study or be using one of the following acceptable birth control methods:

  1. non-hormone releasing intrauterine device in place for at least 3 months prior to the first dose with a physical (e.g. condom or diaphragm or other) and a chemical barrier (e.g. spermicide) from the time of screening through 14 days following the last dose
  2. double physical barrier (e.g. condom and diaphragm or other) and a chemical barrier (e.g. spermicide) from the time of screening through 14 days following the last dose
  3. surgical sterilization of the partner (vasectomy for 180 days minimum) with a physical (e.g. condom or diaphragm or other) and a chemical barrier (e.g. spermicide) from the time of screening through 14 days following the last dose.
  4. or have an exclusive non-heterosexual lifestyle
* In addition, female subjects of childbearing potential will be advised to remain sexually inactive or to keep the same birth control method for at least 14 days following the last dose
* Female of non childbearing potential: must have undergone one of the following sterilization procedures at least 6 months prior to the first dose:

  1. hysteroscopy sterilization (with a copy of the confirmation test) and be using a physical (e.g. condom or diaphragm or other) and a chemical barrier (e.g. spermicide) a barrier method (e.g., condom or diaphragm) with spermicide throughout the study
  2. bilateral tubal ligation or bilateral salpingectomy and be using a physical (e.g. condom or diaphragm or other) and a chemical barrier (e.g. spermicide) a barrier method (e.g., condom or diaphragm) with spermicide throughout the study
  3. hysterectomy
  4. bilateral oophorectomy or be postmenopausal with amenorrhea for at least 1 year prior to the first dose and FSH serum levels consistent with postmenopausal status
* A non vasectomized, male subject must agree to use a condom with spermicide or abstain from sexual intercourse during the study until 90 days beyond the last dose of study drug. (No restrictions are required for a vasectomized male provided his vasectomy has been performed 4 months or more prior to study start. A male who has been vasectomized less than 4 months prior to study start must follow the same restrictions as a non vasectomized male)
* If male, must agree not to donate sperm from the first dose until 90 days after dosing
* A subject who claims to be sexually inactive needs to remain inactive for the whole study duration
* Understands the study procedures in the informed consent form (ICF), and be willing and able to comply with the protocol

Exclusion Criteria:

* Subject is mentally or legally incapacitated or has significant emotional problems at the time of screening visit or expected during the conduct of the study
* History or presence of clinically significant medical or psychiatric condition or disease in the opinion of the PI
* History of any illness that, in the opinion of the PI, might confound the results of the study or poses an additional risk to the subject by their participation in the study
* History or presence of chronic alcohol or drug abuse the past 2 years prior to screening
* History or presence of hypersensitivity or idiosyncratic reaction to the study drug(s) or related compounds (e.g., any other benzodiazepine for midazolam since cross sensitivity with other benzodiazepines is possible) or any component of the midazolam solution formulation
* Subject is currently taking or has a history of pronounced sedation upon taking benzodiazepines or other sedative/soporific drugs
* Female subjects who are pregnant or lactating
* Positive urine drug results at screening or check-in or positive alcohol results at check in
* Drink alcohol in excess of 21 glasses/units per week for males or 14 glasses/units per week for females, with one unit = 150 mL of wine or 360 mL of beer or 45 mL of 45% alcohol
* Positive urine cotinine at screening
* Positive results at screening for HIV, HBsAg or HCV
* Seated blood pressure is less than 90/40 mmHg or greater than 140/90 mmHg at screening
* Seated heart rate is lower than 40 bpm or higher than 99 bpm at screening
* QTcF interval is >430 msec (males) or >450 msec (females) or deemed clinically abnormal by the PI
* Unable to refrain from or anticipates the use of:

  * Any drug, including prescription and non prescription medications, herbal remedies, or vitamin supplements beginning 14 days prior to the first dose of study drug and throughout the study. Hormonal contraceptives and hormone replacement therapy will not be allowed. Paracetamol (up to 2 g per 24 hour period) may be permitted during the study.
  * Any drugs, foods, or herbal preparations known to be significant inducers of CYP enzymes and/or Pgp, including St. John's Wort, for 28 days prior to the first dose of study drug and throughout the study. Appropriate sources will be consulted by the PI or designee to confirm lack of PK/PD interaction with study drug.
* Have been on a diet incompatible with the on study diet, in the opinion of the PI, within the 28 days prior to the first dose of study drug(s), and throughout the study
* Donation of blood or plasma within 90 days prior to the first dose of study drug
* Donation of bone marrow within the last 6 months prior to the first dose of study drug
* Participation in another clinical trial within 90 days prior to the first dose of study drug. The 90 day window will be derived from the date of the last study scheduled blood collection

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2014-09; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
To evaluate the change in maximum plasma concentration (Cmax) and area under the curve (AUC) for both midazolam and 1-OH-midazolam after 7 days of treatment with CTX-4430 | 10 days

SECONDARY OUTCOMES:
To evaluate the safety and tolerability of the administration of single oral doses of midazolam, both in the absence and presence of multiple dose CTX-4430. | 10 days
  Safety and tolerability assessments include Adverse Event monitoring, Physical Examinations, Vital Sign assessments (heart rate, blood pressure, respiratory rate and temperature), Pulse Oximetry assessments, ECG assessments and Pregnancy testing in female subjects.
To evaluate the safety and tolerability of multiple oral doses of CTX-4430. | 10 days
  Safety and tolerability assessments include Adverse Event monitoring, Physical Examinations, Vital Sign assessments (heart rate, blood pressure, respiratory rate and temperature), Pulse Oximetry assessments, ECG assessments and Pregnancy testing in female subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Johnston Stewart, MB, BSc, Principal Investigator — Celerion Belfast, Northern Ireland
Locations (1):
- Celerion, Belfast, United Kingdom